CLINICAL TRIAL: NCT01989741
Title: Effect of Sleep Restriction on Decision Making and Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche Biomedicale des Armees (Other Government)
Responsible Party: Principal Investigator, SAUVET Fabien, médecin principal (MD, PhD), Institut de Recherche Biomedicale des Armees
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2012-A00399-34
Record Dates: First submitted 2013-01-12; First posted 2013-11-21 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Sleep Deprivation
Keywords: sleep restriction, decision making, wakefullness
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sleep restriction (Other): Longitudinal study of response to sleep restriction. Comparison between baseline values and sleep restriction values
  Interventions: Other: Sleep restriction

INTERVENTIONS:
Other: Sleep restriction — 4 hours sleep by night during one week

SUMMARY:
* hypothesis: sleep restriction in healthy subject trigger alteration of decision making associated with immuno-inflammatory changes
* inclusion criterias: healthy subjects, men, under 35 years, BMI<26, no sleep troubles, intermediate chronotype
* design: 12 subjects, longitudinal study 2 days of baseline, 7 night of sleep restriction (4h sleep/night), recovery (1, 2, 3 and 9 normal sleep nights).
* parameters: decision making tests, reaction time, wakefulness test, biological parameters (cathecholamines, pro-inflammatory cytokines...), heart rate, blood pressure
* control of sleep restriction: continuous polysomnographic survey

ELIGIBILITY:
Inclusion Criteria:

* healthy men, < 35 yr old, BMI<26, intermediate chronotype

Exclusion Criteria:

* sleep trouble, acute or chronique disease (cardiological, neurological...), women

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
London tower test score (décision making) | up to 3 days
  % of good score and mean response time resulting from London Tower test, assessed during baseline, sleep restriction (day 1 to day 5) and recovery (day 1 to day 3) at 10 AM

SECONDARY OUTCOMES:
wakefulness | maintenance of wakefulness test (MWT) score observed every day during baselline, sleep restriction and recovery at 09 AM, 12 AM, 4 PM and 7 PM
cognitive function | up to 3 days
Inflammation | biological marker of inflammation levels assessed every day during baseline, sleep restriction and recovery at 08 AM

CONTACTS AND LOCATIONS:
Overall Officials: Fabien SAUVET, MD, PhD, Principal Investigator — Institut de recherche biomédicale des armées
Locations (1):
- Institut de recherche biomédicale des armées, Brétigny-sur-Orge, France

REFERENCES:
- [Derived] Rabat A, Gomez-Merino D, Roca-Paixao L, Bougard C, Van Beers P, Dispersyn G, Guillard M, Bourrilhon C, Drogou C, Arnal PJ, Sauvet F, Leger D, Chennaoui M. Differential Kinetics in Alteration and Recovery of Cognitive Processes from a Chronic Sleep Restriction in Young Healthy Men. Front Behav Neurosci. 2016 May 23;10:95. doi: 10.3389/fnbeh.2016.00095. eCollection 2016. PMID 27242464
- [Derived] Sauvet F, Drogou C, Bougard C, Arnal PJ, Dispersyn G, Bourrilhon C, Rabat A, Van Beers P, Gomez-Merino D, Faraut B, Leger D, Chennaoui M. Vascular response to 1 week of sleep restriction in healthy subjects. A metabolic response? Int J Cardiol. 2015;190:246-55. doi: 10.1016/j.ijcard.2015.04.119. Epub 2015 Apr 16. PMID 25932797